CLINICAL TRIAL: NCT03233256
Title: Rapid Measurements of Water Isotopes in Human Breath and Saliva for Doubly Labeled Water Analysis
Brief Title: Measurements of Water in Breath and Saliva
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-2203; R21DK113401 (NIH)
Record Dates: First submitted 2017-07-25; First posted 2017-07-28 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Human Energy Expenditure

STUDY DESIGN:
Intervention Model Description: Healthy adults (18-45 yrs.) will be recruited from the local Denver area. The investigators have elected to study a relatively homogenous sample to limit the impact of age, weight, and chronic disease on isotope fractionation in breath.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy adults (18-45 yrs.) (Experimental): Healthy adults (18-45 yrs.) will be recruited from the local Denver area. The investigators have elected to study a relatively homogenous sample to limit the impact of age, weight, and chronic disease on isotope fractionation in breath.
  Interventions: Procedure: Feasibility of measuring 2H:1H and 18O:16O in saliva and breath.

INTERVENTIONS:
Procedure: Feasibility of measuring 2H:1H and 18O:16O in saliva and breath. — The investigators propose to demonstrate the feasibility of measuring 2H:1H and 18O:16O in saliva and breath. The natural abundances of 2H:1H and 18O:16O of urine, saliva, and breath samples will be determined from samples obtained simultaneously from 50 relatively healthy human subjects. We will also measure 2H:1H and 18O:16O enrichments in urine, saliva, and breath of 10 relatively healthy human subjects obtained after consuming a standard DLW dose and compare the estimates of TDEE using these different matrices.

SUMMARY:
This study proposes to demonstrate the feasibility of measuring 2H:1H and 18O:16O in saliva and breath by comparing the natural abundances of 2H:1H and 18O:16O in saliva and urine of un-dosed humans.

DETAILED DESCRIPTION:
The scientific premises for this line of research are 1) challenges related to costs, the complexity of sample collection and preparation, and the level of technical skills required for Isotope-ratio mass spectrometry (IRMS) analysis have limited the adoption of the doubly labeled water (DLW) method; and 2) the investigators preliminary data demonstrates that Off-Axis Integrated Cavity Output Spectroscopy (OA-ICOS) provides a valid, more rapid, and less technically challenging approach to isotopic analysis of human samples.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult men and women, aged 18-45 yrs

Exclusion Criteria:

* Obesity (body mass index (BMI) > 30 kg/m2)
* Pregnant or lactating women
* Self-reported acute or chronic disease (diabetes, heart diseases, thyroid diseases)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-02-27 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Natural abundances of 2H:1H and 18O:16O in humans | Baseline
  Evaluation of the natural abundances of 2H:1H and 18O:16O in urine, saliva, and breath of humans.

CONTACTS AND LOCATIONS:
Overall Officials: Edward L Melanson, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Edward Melanson, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No